CLINICAL TRIAL: NCT00756158
Title: Molecular Studies on the Candidate Genes of Dopaminergic and Noradrenergic Systems in Attention-deficit Hyperactivity Disorder
Brief Title: Molecular Studies on the Candidate Genes of Dopaminergic and Noradrenergic Systems in ADHD
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 200712085R
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; dopaminergic; noradrenergic; endophenotype; molecular genetics; candidate gene; Family-based Association study
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Biospecimen Retention: Samples With DNA — The subjects will receive blood withdrawal. The blood sample will be used for establishing lymphoblastoid cell lines, which will be used for molecular genetic experiments
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The ultimate goal of this study is to find specific polymorphism of candidate genes associated with endophenotypes and/or phenomenological phenotypes of ADHD. We propose to replicate the analysis of the candidate genes identified by previous genetic studies on ADHD using the candidate gene association study design (family-based case control study using parental controls) to validate the findings from other research groups. These results will lead our team: (1) to resolve controversies over inconsistent findings in previous genetic studies and contribute to the literature on the validity of ASD using clinical and genetic data; (2) to study the pathogenetic process of abnormal genes in abnormal neuropsychological and neurobiological functions of ADHD; (3) to delineate the nature and the effect of gene-gene interaction in the etiology of ADHD.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD), characterized by inattention, hyperactivity and impulsivity, is an early onset, highly heritable, clinically heterogeneous, long-term impairing disorder with tremendous impact on individuals, families, and societies. It affects 5-10% of school-aged children worldwide (7.5% in Taiwan) and 2-4% of adults. Neuropsychological deficits related to executive functions, state regulation, and delay aversion show heritability, replicated association with ADHD, and familial-genetic overlap with ADHD, are suitable for biomarkers for ADHD. Despite the abundance of molecular genetic studies on ADHD, the genetic etiologies of ADHD have been non-conclusive, and there is limited information about the expressions, neuropsychological deficits, and genetic variants for ADHD in Chinese population. This present study, a family-based parental control association study, aims to identify the genetic markers of dopaminergic and noradrenergic systems for ADHD using the dichotomous categorization of affected and non-affected, quantitative phenotypes (symptom dimension and severity of ADHD) and endophenotype (neuropsychological measures) as well.

Specific Aims:

1. to determine the components of ADHD and neuropsychological deficits with the greatest familial recurrence risks;
2. to replicate studies with positive genetic findings from literature by performing candidate gene analysis such as DRD4, DRD2, DRD5, DAT1, DBH, ADRA2C, ADRA1C, and SLC6A2;
3. to identify the potential genetic variants using haplotype tagSNPs for the following candidate genes, MAO-A and ADRA2A and any updated genetic findings.

In addition to a sample of 200 ADHD families (200 probands, 400 parents, and 150 siblings) being recruited in a parallel study (NSC96-2628-B-002-069 -MY3), we will recruit another 100 probands with ADHD, aged 7-18, and their parents (n = 200) and siblings (n= 75) in this project. The phenotype measures include (1) interviews for psychopathology (K-SADS-E) and social functioning (SAICA), (2) self-administered questionnaires to measures ADHD symptoms (SNAP-IV and Adult ADHD rating scale) and comorbid conditions (ASRI and CBCL), and (3) Neuropsychological tests: WISC-III, CPT, CANTAB, and Time Perception Tasks. The DNA will be collected and analyzed. The transmission/disequilibrium test (TDT) and quantitative TDT will be used in data analysis.

We anticipate the establishment of clinical, neuropsychological, and genetic database of 300 ADHD families (200 in NSC96-2628-B-002-069-MY3 and 100 in this project), completion of the screening of several candidate genes, and identification of potential genetic variants for ADHD, and determination of their association with ADHD diagnosis and symptoms and its endophenotype in a Taiwanese sample. The long-term objectives are to identify the behavioral phenotypes and endophenotypes that are close to the biological expression of genes underlying ADHD. The findings of different approaches to identify the genetic etiologies for ADHD in this pilot study should help us to determine the most promising approach for future molecular genetic and pharmacogenetic study on ADHD.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the proband subjects are
* That subjects have a clinical diagnosis of ADHD, or Hyperkinetic Disorder defined by the DSM-IV and ICD-10, respectively, which was made by a full-time board-certificated child psychiatrist at the first visit and following visits;
* Their ages range from 7 to 18 when we conduct the study;
* Subjects have at least one biological parent;
* Both parents are Han Chinese;
* Subjects and their biological parents (and siblings if any) consent to participate in this study for complete phenotype assessments and blood withdraw or saliva collection for genetic study.

Exclusion Criteria:

* The proband subjects will be excluded from the study if they currently meet criteria or have a history of the following condition as defined by DSM-IV:

  * Schizophrenia,
  * Schizoaffective Disorder,
  * Organic Psychosis, or Pervasive Developmental Disorder.
* Moreover, the subjects will also be excluded from the study if they completely cannot cooperate with blood withdrawal, collection of saliva, or buccal swabs.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The sample will consist of 100 probands with ADHD, aged 7-18. Their biological parents (n = 200) and siblings (estimated number = 75) born to the same biological parents will be recruited as the parent controls and sibling controls, respectively, for the family-based case control study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-08-01 (Actual); Primary Completion 2011-07-31 (Actual); Study Completion 2011-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Yung Shang, MD, Principal Investigator — Dept of Psychiatry, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan